CLINICAL TRIAL: NCT02306863
Title: The Efficacy of Long-term Whole-body Vibration in the Treatment of Parkinson's Disease
Brief Title: Whole-body Vibration as a Treatment for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Adam Koebel, Undergraduate Thesis Student, Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4291
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Parkinson's Disease; Primary Parkinsonism
Keywords: Parkinson's Disease; whole-body vibration; WBV
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- whole-body vibration (Experimental): 40 Hz Whole-body vibration applied via physioaccoustic method for 12 weeks, 3 times a week
  Interventions: Device: vibrating chair
- sham treatment (Sham Comparator): simulated whole-body vibration applied 3 times a week for 12 weeks
  Interventions: Device: sham treatment

INTERVENTIONS:
Device: vibrating chair — vibration provided via physioacoustic method
  Arms: whole-body vibration
Device: sham treatment — simulated whole-body vibration
  Other Names: placebo
  Arms: sham treatment

SUMMARY:
This study will evaluate whether whole-body vibration applied over a 12-week period is effective in treating motor symptoms of Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disease resulting in the loss of dopaminergic neurons projecting from the substantia nigra pars compacta to the striatum.

Whole-body vibration (WBV) is potentially beneficial in treating Parkinson's disease because it has been shown to elicit effects specific to both the brain and muscular system. Animal models of PD indicate that whole-body vibration can increase striatal dopamine levels, as well as the number of dopaminergic neurons in the substantia nigra. These findings were correlated with increased levels of brain-derived neurotrophic factor.

In addition to the potentially neuroplastic effects, >20 Hz WBV has been shown to improve muscular performance. Improved muscular performance is believed to be attributed to WBV induced neuromuscular effects rather than muscle hypertrophy, with the specific mechanism defined as the tonic vibration reflex.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's Disease by a Neurologist
* Currently taking anti-Parkinsonian medication
* Able to stand for 2 minutes without assistance
* Able to walk 10 meters without assistance
* Ability to understand English instructions
* Normal or corrected vision

Exclusion Criteria:

* A neurological disease other than PD
* recent stroke
* cardiovascular disease
* previous major hemorrhage
* artificial pacemaker
* currently pregnant
* Current participation in any physical therapy or experimental treatments
* Peripheral neuropathy, severe osteoporosis
* Visual impairments that cannot be corrected
* Clinically diagnosed with dementia
* Greater than mild dementia (screened using Montreal Cognitive Assessment (MOCA) <24 being excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) section III | change from baseline, 12 weeks, and 2 week washout
  clinician monitored motor evaluation

SECONDARY OUTCOMES:
Gait Assessment | change from baseline, 12 weeks, and 2 week washout
  pressure sensitive carpet (GAITRite) measuring gait parameters (step length, step velocity, stride-to-stride variability, etc)
Timed Up & Go (TUG) Test | change from baseline, 12 weeks, and 2 week washout
  measuring time participants take to stand up from chair, walk towards an obstacle, turn around, walk back to chair, and sit back down again
Timed Grooved Pegboard Task | change from baseline, 12 weeks, and 2 week washout
  25 pegs with a key along one side must be rotated to properly be inserted into slot on board (measuring time-in and time-out)

CONTACTS AND LOCATIONS:
Overall Officials: Adam K Koebel, BSc, Principal Investigator — Wilfrid Laurier University
Locations (1):
- Sun Life Financial Movement Disorders Research & Rehabilitation Centre, Waterloo, Ontario, Canada

REFERENCES:
- [Background] Haas CT, Turbanski S, Kessler K, Schmidtbleicher D. The effects of random whole-body-vibration on motor symptoms in Parkinson's disease. NeuroRehabilitation. 2006;21(1):29-36. PMID 16720935
- [Background] Ebersbach G, Edler D, Kaufhold O, Wissel J. Whole body vibration versus conventional physiotherapy to improve balance and gait in Parkinson's disease. Arch Phys Med Rehabil. 2008 Mar;89(3):399-403. doi: 10.1016/j.apmr.2007.09.031. PMID 18295614
- [Background] King LK, Almeida QJ, Ahonen H. Short-term effects of vibration therapy on motor impairments in Parkinson's disease. NeuroRehabilitation. 2009;25(4):297-306. doi: 10.3233/NRE-2009-0528. PMID 20037223